CLINICAL TRIAL: NCT06431555
Title: Magnetic Resonance Lung Function Imaging Study of Pulmonary Fibrosis Combined With Emphysema Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-ke-107
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-01

CONDITIONS: Using Functional Lung MRI to Explore Pulmonary Perfusion Changes in Patients With Pulmonary Fibrosis and Emphysema Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — Non-contrast, free-breathing MRI scan

SUMMARY:
This study intends to use magnetic resonance pulmonary function imaging technology to explore imaging markers for early diagnosis of patients with CPFE. Through baseline, 6-month and 12-month follow-up examinations, the changes in magnetic resonance pulmonary function in patients with CPFE and their correlation with disease progression were explored.

ELIGIBILITY:
Inclusion Criteria:

* (1) Chest HRCT shows emphysema mainly distributed in the upper lung field, manifesting as wallless or thin-walled (wall thickness <1 mm) low-transmittance areas with clear boundaries with normal tissue, or multiple bullae (diameter > 1 cm), and the emphysema area/total lung volume is ≥10%; (2) interstitial pulmonary fibrosis mainly distributed in the lower lung field and subpleura, manifesting as honeycomb shadow or grid shadow, and the lung structure is destroyed , may be accompanied by traction bronchiectasis, ground glass opacities and consolidation opacities.

Exclusion Criteria:

* (1) Refusal to sign the informed consent form; (2) MRI contraindications (implanted pacemaker/defibrillator, claustrophobia, or any clinical condition that prohibits longer MRI examinations).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: (1) Chest HRCT shows emphysema mainly distributed in the upper lung field, manifesting as wallless or thin-walled (wall thickness <1 mm) low-transmittance areas with clear boundaries with normal tissue, or multiple bullae (diameter > 1 cm), and the emphysema area/total lung volume is ≥10%; (2) interstitial pulmonary fibrosis mainly distributed in the lower lung field and subpleura, manifesting as honeycomb shadow or grid shadow, and the lung structure is destroyed , may be accompanied by traction bronchiectasis, ground glass opacities and consolidation opacities.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
perfusion defect percentage | 12 months
  Calculate MRI lung perfusion defect as a percentage of the whole lung

CONTACTS AND LOCATIONS:
Overall Officials: Shumin Wang, PhD, Study Director — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ouyang T, Wang Y, Zhang H, Voskrebenzev A, Vogel-Claussen J, Ye Q, Yang Q. Ventilation and Perfusion Defects on Phase-Resolved Functional Lung (PREFUL) MRI Predict Silicosis Progression: A Prospective Pilot Study. J Magn Reson Imaging. 2025 Nov 24. doi: 10.1002/jmri.70183. Online ahead of print. PMID 41277498